CLINICAL TRIAL: NCT05970588
Title: Impact of a Standing Desk Converter Intervention on Habitual Posture, Cognition, and Cardiovascular Health
Brief Title: Standing Desk Converter & Habitual Posture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olga Theou (Other)
Responsible Party: Sponsor-Investigator, Olga Theou, Assistant Professor, Dalhousie University
Organization: Dalhousie University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2023-6694
Record Dates: First submitted 2023-07-16; First posted 2023-08-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Sedentary Time; Cognitive Function; Blood Pressure Regulation
Keywords: Standing Time; Occupational Health; Stroop Task; Carotid Intima-Media Thickness; Head-Up Tilt; Objectively Measured Activity
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: A block randomization strategy will be implemented to ensure equal allocations to intervention/control groups in groups of 6 (3 per group). Even and odd numerals will represent designation to the Intervention and Control groups, respectively. For example, if the first 3 participants are randomized to the control group, the next 3 will be allocated to the intervention group. To ensure all control participants will be offered the intervention after their control period, the first 3 participants for the final block of 6 (block 7) will be randomized to the control group first. Randomization will occur after Visit 1 assessments are complete.
Who Masked: Outcomes Assessor
Masking Description: The control group will receive no intervention and will be inherently not blinded to their group allocation. All analyses will be completed by an individual blinded to participants' group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Wait-list Control Group (No Intervention): Fitted with inclinometers/accelerometers at week 0 and week 4 of the intervention period for 7 consecutive days of wear. Measures of cognition and blood pressure regulation will occur at these same timepoints. Daily activities of participants will not be restricted if patients are assigned to the control group.
- Intervention Group (Experimental): Fitted with inclinometers/accelerometers at week 0 and week 4 of the intervention period for 7 consecutive days of wear. Measures of cognition and blood pressure regulation will occur at these same timepoints.
  Interventions: Behavioral: Standing Promotion Intervention

INTERVENTIONS:
Behavioral: Standing Promotion Intervention — Participants will be provided with a standing desk converter to set on top of their existing desk for 4 weeks.
  Arms: Intervention Group

SUMMARY:
This project will determine the short-term impact of a standing desk converter on: 1) objectively measured physical activity and posture levels, and 2) brain (cognition) and heart (blood pressure regulation) function. The main outcome is habitual activity patterns, assessed by the thigh-worn inclinometer (activPAL). All participants will be equipped with an activPAL and have their cardiovascular and cognitive function assessed at baseline and 4 weeks. Participants in the intervention group will use a standing desk converter for 4 weeks, while the wait-list control group will be encouraged to maintain their regular activity patterns. Researchers will compare the intervention and control groups to see if using the standing desk converter will increase standing time and lower sedentary time, improve cognition, and improve blood pressure regulation.

DETAILED DESCRIPTION:
Background: Too much sedentary time (time spent sitting, reclining, or lying) leads to health problems such as cognitive impairments or cardiovascular disease. A lot of sedentary time is accumulated while working at a desk (e.g., computer work, studying, etc.). Standing desk interventions have provided mixed support as to whether they can reduce habitual sedentary time, with the need for more controlled interventional studies. It remains to be determined if a simple standing desk converter (i.e., a height-adjusted desk that can be set on top of a traditional sitting desk) increases standing time (i.e., not sedentary) and/or decreases sedentary time. Worse cognitive health and higher blood pressure are linked to a greater risk of chronic conditions such as dementia and cardiovascular disease, respectively. More physical activity improves cognition and blood pressure regulation, but whether standing more also translates to these brain and heart improvements is unclear.

Main Objective: The goals of this project are to determine the impact of a standing desk converter on: 1) objectively measured physical activity and posture levels, and 2) brain (cognition) and heart (blood pressure regulation) function. It is expected that using the standing desk converter will increase standing time and lower sedentary time, improve cognition, and improve blood pressure regulation.

Methodology: For the proposed project, we will assess free-living posture, cognition, and blood pressure regulation before and after 4-weeks of either using a standing desk converter (intervention) or a wait-list control. The study population targets adults who use a traditional seated desk for a minimum of 20 hours per week and do not already use a standing desk. Free-living activity will be assessed using activity monitors (activPALs) worn for 7-days before and after either the control period or intervention. Cognition will be assessed using a computerized Stroop task that records accuracy and reaction times to selecting the colour of the word or the word itself (e.g., word BLUE written in red font). Progressively more challenging Stroop conditions will be used to assess different aspects of cognition. During the Stroop, cerebral oxygenation will be determined using near-infrared spectroscopy. Beat-by-beat blood pressure (via finger cuff), heart rate (via electrocardiogram), and internal carotid artery size and red blood cell velocity (via ultrasound) will be measured while lying down and in response to 20 minutes of 60-degree passive head-up tilt that tests blood pressure regulation. The proposed study will yield new knowledge as it relates to real-life posture interventions that promote healthier movement and investigates whether standing converters lead to improvements in brain and heart health.

Significance: The proposed study will yield new knowledge as it relates to real-life posture interventions that promote healthier movement and investigates whether standing converters lead to improvements in brain and heart health.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Are normotensive, cognitively healthy, and do not have a history of fainting while standing
* Are able to stand for 10 min without assistance (e.g., require a walker, person assistance)
* Are not allergic to clear medical adhesive (TegadermTM, 3M) used to secure the activPAL activity monitors
* Use a seated desk at least 20 hours/week in the last month and do not use a standing or active desk already
* Females who are not pregnant, breastfeeding or planning on becoming pregnant prior to entry into the study

Exclusion Criteria:

* Younger than 18 years old
* Hypertension (resting systolic pressure >139 mmHg and/or diastolic pressure >89 mmHg)
* Have a diagnosed cognitive impairment
* Have a history of orthostatic hypotension/intolerance and/or fainting while standing
* Cannot stand for at least 10 min without assistance (e.g., require a walker, person assistance)
* Have a known allergy to the clear medical adhesive (TegadermTM, 3M)
* Use a seated desk less than 20 hours/week, use a standing or active desk already, or use a desk for more than 20 hours/week but not in the last month
* Females who are pregnant, breastfeeding or planning on becoming pregnant prior to entry into the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
ActivPAL monitors | Change from baseline (week 0) activity to post intervention (week 4).
  Habitual sedentary and physical activity data will be recorded through the thigh-worn monitor. Information obtained from the 3 monitors will provide information regarding time spent lying, sitting (bent vs straight leg) and standing.

SECONDARY OUTCOMES:
Cognition | Change from baseline (week 0) activity to post intervention (week 4).
  The computerized Stroop task will consist of the three conditions mentioned above: simple, interference, and switching. The computer program used to administer the task records accuracy and reaction time.
Brain Activation: Functional Near Infrared Spectroscopy | Change from baseline (week 0) activity to post intervention (week 4).
  Functional Near Infrared Spectroscopy (fNIRS) is a well-established modality of neuroimaging that can detect differences in blood-oxygen-level dependent (BOLD) signal, allowing one to make inferences on brain activity. fNIRS sensors consist of light sources that emit near-infrared light, as well as photo diodes that detect the levels of the light at the two different frequencies. As each wavelength of light is known to be absorbed differently by oxy- and deoxyhemoglobin, one can infer cerebral oxygenation via the relative absorption of each wavelength through the application of a modified beer-lambert law. The NIRScout system contains 8 LED sources and 16 detectors (optodes), which can be placed in customized configurations to measure from different regions of the brain. The sources and detectors are held in place through an elasticized cap that fastens with Velcro under the chin.
Electrocardiography | Change from baseline (week 0) activity to post intervention (week 4).
  Heart rate will be monitored via electrocardiography (ECG). ECG is the non-invasive, passive recording of electrical cardiac activity at the surface of the skin. This will be recorded at a sampling frequency using a dedicated data acquisition system (PowerLab, ADInstruments) and analysis software (Lab Chart, ADInstruments).
Continuous Finger Blood Pressure Recording (Finapres Medical Systems) | Change from baseline (week 0) activity to post intervention (week 4).
  A small cuff used to measure continuous, non-invasive blood pressure will be placed around the middle or index finger. When in use, the cuff will inflate with air and gently squeeze the finger. This will be recorded at a sampling rate of 200Hz using a dedicated data acquisition system (PowerLab, ADInstruments) and analysis software (Lab Chart, ADInstruments).
Upper Arm Blood Pressure Measurements | Change from baseline (week 0) activity to post intervention (week 4).
  A semi-automated patient vital signs monitor (Carescape v100®, General Electric Healthcare) will be used to record resting, seated blood pressure from the upper left arm (i.e., the brachial artery). Additional measurements will be recorded during the various rest periods.
Carotid Artery Structure | Change from baseline (week 0) activity to post intervention (week 4).
  Internal carotid artery intima-media thickness will be imaged on the right-side. A minimum of two minutes of beat-by-beat carotid images during supine rest, the initial tilt, and the final tilt period will be collected.
Carotid Artery Function | Change from baseline (week 0) activity to post intervention (week 4).
  Internal carotid artery function changes in blood flow to head-up tilt will be measured via ultrasonography. A minimum of two minutes of beat-by-beat carotid images during supine rest, the initial tilt, and the final tilt period will be collected in the right-side common carotid artery.

CONTACTS AND LOCATIONS:
Overall Officials: Myles W O'Brien, PhD, Principal Investigator — Department of Medicine and Department of Physiotherapy, Dalhousie University
Locations (1):
- Dalhousie University, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dorey TW, O'Brien MW, Robinson SA, Kimmerly DS. Knee-high compression socks minimize head-up tilt-induced cerebral and cardiovascular responses following dynamic exercise. Scand J Med Sci Sports. 2018 Jul;28(7):1766-1774. doi: 10.1111/sms.13084. Epub 2018 Apr 16. PMID 29575406
- [Background] Neuhaus M, Eakin EG, Straker L, Owen N, Dunstan DW, Reid N, Healy GN. Reducing occupational sedentary time: a systematic review and meta-analysis of evidence on activity-permissive workstations. Obes Rev. 2014 Oct;15(10):822-38. doi: 10.1111/obr.12201. Epub 2014 Jul 11. PMID 25040784
- [Background] O'Brien MW, Daley WS, Schwartz BD, Shivgulam ME, Wu Y, Kimmerly DS, Frayne RJ. Characterization of Detailed Sedentary Postures Using a Tri-Monitor ActivPAL Configuration in Free-Living Conditions. Sensors (Basel). 2023 Jan 4;23(2):587. doi: 10.3390/s23020587. PMID 36679384
- [Background] Petterson, JL, Mekari, S, O'Brien, MW. An open-source Stroop task program that incorporates a switching condition to determine executive function. Software Impacts. 2022 Jul 7 13, 100361. doi: 10.1016/j.simpa.2022.100361
- [Background] de Rezende LF, Rodrigues Lopes M, Rey-Lopez JP, Matsudo VK, Luiz Odo C. Sedentary behavior and health outcomes: an overview of systematic reviews. PLoS One. 2014 Aug 21;9(8):e105620. doi: 10.1371/journal.pone.0105620. eCollection 2014. PMID 25144686
- [Background] Thorp AA, Healy GN, Winkler E, Clark BK, Gardiner PA, Owen N, Dunstan DW. Prolonged sedentary time and physical activity in workplace and non-work contexts: a cross-sectional study of office, customer service and call centre employees. Int J Behav Nutr Phys Act. 2012 Oct 26;9:128. doi: 10.1186/1479-5868-9-128. PMID 23101767
- [Background] O'Brien MW, Kimmerly DS, Mekari S. Greater habitual moderate-to-vigorous physical activity is associated with better executive function and higher prefrontal oxygenation in older adults. Geroscience. 2021 Dec;43(6):2707-2718. doi: 10.1007/s11357-021-00391-5. Epub 2021 Jun 3. PMID 34081258
- [Background] De Vries J, Michielsen HJ, Van Heck GL. Assessment of fatigue among working people: a comparison of six questionnaires. Occup Environ Med. 2003 Jun;60 Suppl 1(Suppl 1):i10-5. doi: 10.1136/oem.60.suppl_1.i10. PMID 12782741
- [Background] Hatoum T, Sheldon R. A practical approach to investigation of syncope. Can J Cardiol. 2014 Jun;30(6):671-4. doi: 10.1016/j.cjca.2014.03.043. Epub 2014 Apr 3. PMID 24882540
- [Background] Petersen ME, Williams TR, Gordon C, Chamberlain-Webber R, Sutton R. The normal response to prolonged passive head up tilt testing. Heart. 2000 Nov;84(5):509-14. doi: 10.1136/heart.84.5.509. PMID 11040011
- [Background] Bantoft C, Summers MJ, Tranent PJ, Palmer MA, Cooley PD, Pedersen SJ. Effect of Standing or Walking at a Workstation on Cognitive Function: A Randomized Counterbalanced Trial. Hum Factors. 2016 Feb;58(1):140-9. doi: 10.1177/0018720815605446. Epub 2015 Sep 24. PMID 26408647
- [Background] E F Graves L, C Murphy R, Shepherd SO, Cabot J, Hopkins ND. Evaluation of sit-stand workstations in an office setting: a randomised controlled trial. BMC Public Health. 2015 Nov 19;15:1145. doi: 10.1186/s12889-015-2469-8. PMID 26584856
- [Background] Ma J, Ma D, Li Z, Kim H. Effects of a Workplace Sit-Stand Desk Intervention on Health and Productivity. Int J Environ Res Public Health. 2021 Nov 4;18(21):11604. doi: 10.3390/ijerph182111604. PMID 34770116